CLINICAL TRIAL: NCT04306523
Title: Early Genetic and Environmental Influences on Eating: The Baylor Infant Twin Study (BITS)
Brief Title: Early Genetic and Environmental Influences on Eating - The Baylor Infant Twins Study
Acronym: BITS
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Alexis Wood, Assistant Professor, Baylor College of Medicine
Other Study IDs: H-36097
Record Dates: First submitted 2020-01-30; First posted 2020-03-13 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Body Composition; Executive Functioning; Temperament
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — infant: urine sample, fecal sample, fingernails, buccal /saliva sample maternal: buccal sample, saliva sample, fecal sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational Cohort: One group of 100 sets of twin infants, observed from 4 months of age until 2years of age.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — 4 months: observation of infant feeding behavior, behavior/temperament; bio-specimen collection; body composition, sucking intensity/frequency, activity intensity/frequency; maternal reports of feeding and behavior/temperament; maternal biospecimen. 6 month: behavior/temperament assessment, physical activity, and body composition. 12 month: Feeding behavior, behavior/temperament assessment, physical activity, and body composition. 24 month: maternal reports of children's eating behavior, behavior/temperament.

SUMMARY:
The purpose of this study is to better understand the genetic and environmental etiology of early infant effortful control and infant feeding behaviors, and preschool executive functioning and eating behaviors. An additional purpose is to establish whether these four constructs (infant effortful control; infant feeding behaviors; preschool executive functioning; and preschool eating behaviors) have shared genetic and / or environment etiologies.

Study objectives:

(1) Evaluate the extent to which genetic influences on infants' effortful control of behavior are modified by prenatal diet, exercise and stress (2) Estimate the extent to which infant effortful control of behavior predicts and shares genetic influences with preschool executive functioning, and preschool eating behaviors. (3) Identify which genes are associated with infant effortful control behavior, preschool executive functioning, and preschool eating behaviors. (4) Examine whether there is a pattern of bacteria in the gut microbiome which associates with infant effortful control of behavior, preschool executive functioning, and preschool eating behaviors.

DETAILED DESCRIPTION:
The Baylor Infant Twin Study will conduct data collection at four time points. Three visits will occur at the Children's Nutrition Research Center (CNRC) Metabolic Research Unit at 4 months, 6 months and 12 months. At 4 and 6 months of age, a home visit will also be conducted. At 24 months of age, study related questionnaires will be sent by postal mail to be completed and returned to research study staff.

Details of each visit:

4 months: Mother and twin infants will be admitted to the Children's Nutrition Research Center (CNRC) Metabolic Research Unit (MRU) at four months corrected gestational age, written consent will be obtained. At the initial visit, procedures for each infant and mother will be completed. For each infant, the procedures to be completed at 4 months will be (1) an observation of the infant's feeding; for this procedure, while the mother is feeding a infant his/her formula or breast milk(bottle or by breast), a video camera will be recording the session. If needed, research staff will coordinate timing so that the infants are fed so that one follows the other. On the other hand, if the infants are usually fed together (tandem feeding of twin infants), the feeding bottles (or nursing at breast) will be given to each infant at the same time and mother will feed twin infants together during the feeding episode as she normally would do. (2) During the feeding episode, for infants who are being bottle fed, the mother will be asked to use an ordinary infant feeding bottle with an added special pressure sensor while infant sucks their regular feed from it. The device is a regular baby bottle that has a special pressure sensing chamber that measures the infant's sucking patterns, strength and consistency. The mother may decline using the bottle with sensors, or if tried with the infant but the infant refuses, the feeding will be resumed with the bottle brought by the mother. (3) Body composition of the infant will be measured using Dual-Energy X-Ray Absorptiometry (DXA) using a Hologic Delphi-A densitometer. These procedures provide estimates of total body bone, fat, and lean mass. (4) Observations of infant's behavior will be observed and recorded for 20 minutes in these situations: being shown a black and white checkerboard, listening to a ringing bell, listening and viewing a shaken ball/rattle, and being presented a ball/rattle, that is later taken away, a puppet game, peek-a-boo game, playing in a jungle gym, and infant viewing pictures on a computer screen. (5) The physical activity of the infant will be measured for about 1.5 hours by using three ActiGraph GT3X+ accelerometers (Pensacola, FL, USA), placed on each leg of the infant (below knee and above the ankle), another device on the infant's waist. (6) A microbiome sample from the infant will be obtained by study staff collecting fecal sample from diaper for the pattern of bacteria in infant's gut. (7) A urine sample will be obtained for epigenetic (methylation) analysis and will be collected by using a special bag that will be placed over the infant's genital area. (8) Finger nail samples will be obtained by gentle clipping for epigenetic (methylation) analysis. (9) A saliva sample for genetic DNA analysis will be collected. To collect the saliva sample, a staff member will gently rub a stick with a cotton end (similar to a Q-tip) against the infant's cheek for about 30 seconds.

The mother will be asked to complete questionnaires for each infant: Infant Behavior Questionnaire - Very Short Version, Milestones Questionnaire, Infant Feeding History Questionnaire, and Infant Eating Behavior Questionnaire. The mother will be asked to complete procedures at the initial visit. First, a maternal microbiome sample; the mother will be instructed how to collect her fecal sample in the MRU or at her home. Second, a maternal buccal cell sample will be collected from the mother by gently rubbing a stick with a cotton end (similar to a Q-tip) against mother's cheek for about 30 seconds. The mother will be asked to collect her own saliva in a container provided to her.

Home visit: Within a week a home visit will be scheduled to assess infants' behavior. The same process conducted in the laboratory will be conducted at home where infant's behavior will be observed and recorded for 20 minutes in these situations: being shown a black and white checkerboard, listening to a ringing bell, listening and viewing a shaken ball/rattle, and being presented a ball/rattle, that is later taken away, a puppet game, peek-a-boo game, playing in a jungle gym, and baby viewing pictures on a computer screen.

6 months: Behavior observation, physical activity and body composition measurement outlined above will be conducted. The mother will complete Infant Behavior Questionnaire - Very Short Version, Milestones Questionnaire, Infant Feeding History Questionnaire, and Infant Eating Behavior Questionnaire.

Home visit: Within a week a home visit will be scheduled to assess infants' behavior as outlined above.

12 months: Behavior observation, physical activity, body composition measurement outlined above will be conducted. Additionally, a feeding observation to asses food neophobia in twins will be conducted. The mother will be asked to offer a new food (Quinoa or Couscous) to the infant. Infant's response to the new food will be video recorded for 3 minutes. The mother will complete Infant Behavior Questionnaire - Very Short Version and Child Eating Behavior Questionnaire (CEBQ).

24 month: Mother will be sent (via mail) four Questionnaires for each child: Strength and Difficulty Questionnaire (SDQ), Milestone Questionnaire, Eating Behavior (Children's Eating Behavior Questionnaire (CEBQ)), Height And Weight Questionnaire. All questionnaires will be mailed and when completed the mother will return to research staff in a self-addressed envelope.

ELIGIBILITY:
Inclusion Criteria:

Infants from a multiple pregnancy (twins only)

* Born at > 34 weeks gestation,
* Not less than 1800 grams birth weight
* No diagnosis of twin to twin transfusion syndrome, or intrauterine growth retardation

Exclusion Criteria:

* Singleton infant
* Gestational less than 34 weeks
* Birthweight less than 1800 grams
* Diagnosis of twin to twin transfusion syndrome, or intrauterine growth retardation

Ages: 4 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Twin infants
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2015-10; Primary Completion 2024-07 (Actual); Study Completion 2024-07 (Actual)

PRIMARY OUTCOMES:
Infant Behavior Questionnaire (IBQ) | 4 months
  IBQ is a mother-reported Infant temperament scale comprised of 37 items that measure the frequency of range of specified infant behaviors over the last two weeks that assess three aspects of temperament 1. Positive affectivity/surgency (PAS), 2. Negative emotionality (NEG), and 3. Orienting and regulatory capacity (ORC) on a scale ranging from 1-7. A higher score indicates a higher frequency of behavior and a lower score indicates a lower frequency of the behavior.
Infant Behavior Questionnaire (IBQ) | 6 months
  IBQ is a mother-reported Infant temperament scale comprised of 37 items that measure the frequency of range of specified infant behaviors over the last two weeks that assess three aspects of temperament 1. Positive affectivity/surgency (PAS), 2. Negative emotionality (NEG), and 3. Orienting and regulatory capacity (ORC) on a scale ranging from 1-7. A higher score indicates a higher frequency of behavior and a lower score indicates a lower frequency of the behavior.
Infant Behavior Questionnaire (IBQ) | 12 months
  IBQ is a mother-reported Infant temperament scale comprised of 37 items that measure the frequency of range of specified infant behaviors over the last two weeks that assess three aspects of temperament 1. Positive affectivity/surgency (PAS), 2. Negative emotionality (NEG), and 3. Orienting and regulatory capacity (ORC) on a scale ranging from 1-7. A higher score indicates a higher frequency of behavior and a lower score indicates a lower frequency of the behavior.
Rejection of novel food | 12 months
  Observer coded food neophobia will be assessed by video recording infant's reaction to a novel food. The coding will be based on the scale developed by, and utilized in, MOding, Birch and Stifter, 2014, Appetite
Child Eating Behavior Questionnaire (CEBQ) | 24 months
  CEBQ is a parent-report measure comprised of 35 items, each rated on a five-point likert scale that ranges from never to always. It is made up of eight eating behavior sub-scales: Food responsiveness, Emotional over-eating, Enjoyment of food, Desire to drink, Satiety responsiveness, Slowness in eating, Emotional under-eating, and Food fussiness. A higher mean score for each specific sub-scale suggest the child shows a higher tendency toward the respective eating behavior. For example a higher mean score on food responsiveness suggests the child is food responsive.
Laboratory Temperament Assessment Battery (Lab-Tab) | 4 months
  Lab-Tab is an assessment of infant temperament using laboratory observations
Laboratory Temperament Assessment Battery (Lab-Tab) | 6 months
  Lab-Tab is an assessment of infant temperament using laboratory observations
Laboratory Temperament Assessment Battery (Lab-Tab) | 12 months
  Lab-Tab is an assessment of infant temperament using laboratory observations

SECONDARY OUTCOMES:
Body composition | 4 months
  Percentage body fat using DXA scan
Body composition | 6 months
  Percentage body fat using DXA scan
Body composition | 12 months
  Percentage body fat using DXA scan
Height | 4 months
  Child's recumbent length in centimeters will be measured
Height | 6 months
  Child's recumbent length in centimeters will be measured
Height | 12 months
  Child's recumbent length in centimeters will be measured
Weight | 4 months
  Child's weight in kilograms will be measured using digital scale
Weight | 6 months
  Child's weight in kilograms will be measured using digital scale
Weight | 12 months
  Child's weight in kilograms will be measured using digital scale
Microbiome analysis of fecal samples from infant, child, and mother | 4 months
  The bacterial pattern of the infant, child's, and maternal samples of stool will be assayed.
Genetic and Epigenetic analyses of selected genes | 12 months
  The presence of selected genes related to effortful control, executive functioning, and eating behavior will be assayed from saliva and buccal samples; The epigenetic (methylation) status of selected genes will be compared in urine and fingernail samples of infants.

CONTACTS AND LOCATIONS:
Overall Officials: Alexis C Wood, PhD, Principal Investigator — Children's Nutrition Research Center, Baylor College of Medicine
Locations (1):
- Children's Nutrition Research Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No data of individuals will be shared